CLINICAL TRIAL: NCT04756921
Title: Pretreatment 18F-FDG Uptake Heterogeneity Predicts Response to Pyrotinib in Patients With Metastatic HER2-positive Breast Cancer
Brief Title: 18F-FDG Uptake Heterogeneity Predicts Pyrotinib Response
Status: Completed | Type: Observational
Sponsor: Biyun Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Biyun Wang, MD, Clinical Professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: YOUNGBC-13
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients cohort: Patients with HER2 positive MBC in the Fudan University Shanghai Cancer Center who underwent whole-body 18F-FDG PET/CT before the initiation of pyrotinib was included.
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400mg po qd

SUMMARY:
Heterogeneity of 18F-fluorodeoxyglucose (FDG) uptake is a promising marker for predicting response to treatment. This study aimed to evaluate the ability of pretreatment positron emission tomography/computed tomography (PET/CT) 18F-FDG-based heterogeneity to predict the response to pyrotinib in patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HER2 positive breast cancer
* Treated with Pyrotinib in the metastatic settings
* Underwent whole-body FDG PET/CT within 4 weeks before the initiation of pyrotinib and capecitabine were included in this study

Exclusion Criteria:

* Incomplete medical history
* Loss of follow up

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HER2 positive breast cancer with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
PFS | Through study completion, an expected average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China